CLINICAL TRIAL: NCT06074250
Title: Targeting Maternal Gut to Improve Mental Health Outcomes-- A Feasibility Pilot Clinical Trial
Brief Title: Perinatal Depression & Anxiety (PDA) and Maternal Gut Microbiome
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Lotte & John Hecht Memorial Foundation (Other)
Responsible Party: Principal Investigator, Neda Ebrahimi, Head of Microbiome Research, The Canadian College of Naturopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CCNMREB049
Record Dates: First submitted 2023-08-03; First posted 2023-10-10 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Perinatal Depression; PerinatalAnxiety
Keywords: Gut Microbiome; Gut-Brain Axis; Diet; Omega 3 Fatty acids; Probiotics; Fish Oil; Mental Health disorders; Perinatal Depression and anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Fish Oils; Docosahexaenoic Acids; Probiotics; Prebiotics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gutopia (Experimental): Women in this arm will receive dietary modification, fish oil and probiotics from the time of enrollment till completion of last study visit (12 months postpartum). The dietary modification will be conducted by a dietician that will provide feedback on the participants diet at enrollment, ways to improve diet quality to meet pregnancy needs, and increase prebiotic foods. Weekly follow-ups will be conducted by the research team to ensure dietary target is met and to help address challenges in doing so. The initial dietary consult will be 30-45 minutes long with 10-15 minute for each subsequent follow-up.
  Interventions: Dietary Supplement: Fish oil; Dietary Supplement: Probiotics; Behavioral: Prebiotics
- Gutboost (Experimental): Women in this arm will receive a daily probiotic and fish oil supplement from the time of enrollment till 1 year postpartum.
  Interventions: Dietary Supplement: Fish oil; Dietary Supplement: Probiotics
- Gutless (Experimental): Women in this arm will receive fish oil and placebo probiotic from the time enrollment till 1 year postpartum .
  Interventions: Dietary Supplement: Fish oil
- Gutnone (Active Comparator): Women in this arm will only be receiving standard care by their obstetrician, and a one time, 30 minutes consult on how to improve baseline diet quality to meet pregnancy needs will be provided by a dietician at the time of enrollment.
  Interventions: Behavioral: Diet Quality

INTERVENTIONS:
Dietary Supplement: Fish oil — 1500mg EPA +1000mg DHA daily
  Other Names: Ecosapentaenoic Acid (EPA); Docosahexaenoic Acid (DHA)
  Arms: Gutboost; Gutless; Gutopia
Dietary Supplement: Probiotics — Combination strain of lactobacillus and bifidobacteria
  Arms: Gutboost; Gutopia
Behavioral: Prebiotics — Dietary consult with follow-up to ensure target fiber intake is met.
  Arms: Gutopia
Behavioral: Diet Quality — one time dietary consult at enrollment to discuss strategies to improve overall diet.
  Arms: Gutnone

SUMMARY:
Perinatal depression and anxiety (PDA) are the leading causes of maternal mortality in developed countries. Women with a history of depression have a 20 fold higher risk of PDA at subsequent pregnancies. The adverse outcomes extend beyond maternal well-being to long-term deficits in children and families. The gut-brain axis is a newly recognized key player in mental health disorders. Specifically, the microbial composition of the gut along with their metabolites are directly involved in disease onset and course. Recent clinical studies have identified diet as the most powerful environmental factor in manipulating gut microbiome. Given vulnerability and resistance of pregnant women to pharmacotherapy, particularly in those with a predisposition to mood disorders, as well as pregnant women's high motivation and commitment to improving gestational diet, a dietary/supplemental intervention to 'optimize' gut microbiome, is a favored approach in disease management. The study investigators aim to exploit microbial responsiveness to diet together with this maternal motivation, to alter the risk and severity of a universal public health concern that has dire and long-term consequences for new moms and their children.

The investigators of this trial, will first study the challenges in pursuing a study aimed at changing the microbiome of pregnant women with a history of mood disorders. Pregnant women in their second trimester will be recruited. Each will be assigned or randomized to one of four groups that will use a combination of diet, supplementation with probiotics, fish oil or no intervention. Each participant will meet with the study team virtually every 3 months until 1 year after delivery. At each study visit participants will be required to complete some questionnaires about their food intake, mood, and other health related measures and will provide a stool sample using the stool collection kits provided.

The findings from this study will help strategize for a larger study that will allow for comparison of the effects of diet, and/or supplementation with Omega-3 Fatty Acids (O3FA) and probiotics on the microbiome and the onset and severity of PDA.

DETAILED DESCRIPTION:
Pregnant women with a history of anxiety and/or depression & currently stable, will be recruited and randomized or assigned to one of four study groups. A total of 100 will be recruited and required to complete six study visits, one every 3 months. At each visit, data on dietary intake, mental health scores, and stool samples will be collected using appropriate tools. All visits will be completed virtually, unless participants need in-person follow-ups.

The final visit is expected to occur between 9-12 months after delivery. The primary outcome for this study is feasibility, measured by: recruiting the targeted number of participant within the anticipated timeframe, and completion of at least 4 of the 6 visits by each participant.

ELIGIBILITY:
Inclusion Criteria

* Women 18-43 years old
* 12-35 weeks of gestation
* Non-smoker/alcohol/recreational drug user
* Financially stable
* Clinical diagnosis of lifetime depression/anxiety or PDA but currently well
* English speaking

Exclusion Criteria:

* Body Mass Index (BMI)≥30
* Low income (unable to afford basic daily needs (i.e., shelter, food, etc.)
* Diagnosis with other major mental health disorders (Bipolar, Psychosis, Addiction, Schizophrenia);
* Diagnosis with other severe medical conditions (i.e. epilepsy, neurological disorders, etc.)
* Allergies to fish oils/ingredients in supplements
* Conditions that require repeated/chronic antibiotic usage
* Having a child with significant mental/physical disability
* Single mothers without any kind of family support,
* Cigarette, alcohol and recreational drug users
* Women unwilling to switch to study product(s)
* Multiparous women with young children (i.e. one or more children less than 4 years of age at the time of delivery)
* Non-English Readers/Speakers

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of participant recruitment | 20 months
  Time taken to recruit 100 participants in total and successfully randomize/assign 25 participants per study arm.
Adherence to Supplement Intake (estimated using unused portion of supplements) | 2 years
  This outcome will be measured by participants' adherence to the prescribed regiments. At each visit the between-study-visit intake of fish oil, probiotics/ placebo will be
  estimated by what remains unused in the original boxes/containers
Adherence to Supplement Intake (Number of missed doses/week) | 2 years
  Questionnaires detailing intake frequency of the supplements and missed doses will be used in Groups A, B & C, to assess adherence to prescribed regiments
Adherence to Dietary Protocol (Using food frequency questionnaire) | 2 years
  Adherence to the dietary protocol in Group A, will be measured at each study visit and in between study visits to ensure the dietary target is met (i.e. the number of daily servings of specific foods are consumed), and to address and document challenges in reaching the targets.
Completion of Study visits(Number of studies with completed tasks) | 2 years
  At each visit participants are expected to provide (1)dietary intake using myfitnesspal, (2) Mental health Scores using Edinburgh Postnatal Depression Scale (EPDS) and General Anxiety Disorder-7 (GAD-7) scales, (3) one stool sample, and 4)provide update on lifestyle and health status. A study visit will be marked complete, only if all tasks are completed. Our benchmark for success is for at least 4 of the 6 study visits to be completed by each participants

SECONDARY OUTCOMES:
Study Obstacles (descriptive measures outlining obstacles) | 2 years
  The actual rate of recruitment, intervention acceptability, completion of study tasks (Dietary intake, EPDS, GAD6, stool collection, lifestyle questionnaires), study visit (<6 visits) will be compared to the expected rates at the time of study design. All obstacles to attaining the expected rate, will be documented with descriptive measures.

CONTACTS AND LOCATIONS:
Overall Officials: Neda Ebrahimi, PhD, Principal Investigator — Canadian College of Naturopathic Medicine
Locations (1):
- Sunnybrook Health Science Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gallant F, Cooley K, Grigoriadis S, Ebrahimi N. Targeting maternal gut microbiome to improve mental health outcomes-a pilot feasibility trial. Front Psychiatry. 2024 Aug 7;15:1414291. doi: 10.3389/fpsyt.2024.1414291. eCollection 2024. PMID 39171074